CLINICAL TRIAL: NCT05130385
Title: Investigation of Retinal Pathology in Eye Diseases Using High Resolution Optical Coherence Tomography (High-Res-OCT)
Brief Title: High Resolution Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: High Res OCT; 2021-D0038 (Registry Identifier: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2021-10-15; First posted 2021-11-23 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Retinal Disease; Retinal Detachment; Retinal Vein Occlusion; Retinal Dystrophy; Retinal Artery Occlusion; Retinal Edema; Retinal Neovascularization; Uveitis; Diabetic Retinopathy; Diabetic Macular Edema; Macular Edema; Macular Degeneration; Macular Disease; Glaucoma; Optic Nerve Diseases; Hypertensive Retinopathy
Keywords: Optical Coherence Tomography; Diagnostic Techniques, Ophthalmological; High resolution optical coherence tomography
MeSH Terms: conditions — Retinal Diseases; Retinal Detachment; Retinal Vein Occlusion; Retinal Dystrophies; Retinal Artery Occlusion; Papilledema; Retinal Neovascularization; Uveitis; Diabetic Retinopathy; Macular Edema; Macular Degeneration; Glaucoma; Optic Nerve Diseases; Hypertensive Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Diabetic Retinopathy: Patients with various degree of diabetic retinopathy
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Artery and vein occlusion: Patients with history of artery or vein occlusion (central or branch artery)
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Glaucoma: Patients with history of glaucoma (open-angle glaucoma, chronic angle closure glaucoma)
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Optic nerve neuropathy: Patients with history of various optic nerve neuropathies
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Hereditary retinal diseases: Patients with history of various retinal dystrophies
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Retinal detachment: Patients history of retinal detachment
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Age related macular degeneration: Patients with history of age related macular degeneration
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Retinal changes from arterial hypertension: Patients with history of arterial hypertension
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Uveitis: Patients with history of uveitis intermedia and/or posterior and/or pan-uveitis
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)
- Healthy: Healthy age matched control subjects
  Interventions: Device: High-resolution optical coherence tomography (High-Res-OCT); Device: Standard spectral domain OCT (SD-OCT)

INTERVENTIONS:
Device: High-resolution optical coherence tomography (High-Res-OCT) — Imaging with high-resolution optical coherence tomography
Device: Standard spectral domain OCT (SD-OCT) — Imaging with standard spectral domain OCT

SUMMARY:
Comparison of high-resolution optical coherence tomography (High-Res-OCT) to conventional imaging modalities for the diagnosis of eye diseases

DETAILED DESCRIPTION:
The high resolution optical coherence tomography (High-Res-OCT) is an improvement of a non-invasive routinely used imaging technique, the optical coherence tomography (OCT), with a light-source capable of providing an increased axial resolution. The routinely used Spectral-Domain OCT has a center wavelength of 880 nm and a spectral bandwidth of 40 nm, resulting in an axial resolution of approximately 7 μm in the eye and is used routinely worldwide. The High-Res OCT works with a central wavelength of 840 nm and an increased bandwidth of 130 nm, making it possible to improve the optical axial resolution in tissue from 7 to 3 µm, without increasing the maximum laser exposure limit. The improved axial resolution of the High-Res OCT results in clearer and more detailed images. The technique is routinely used in clinical practice and the device used for High-Res-OCT (Heidelberg, SPECTRALIS® High-Res OCT- DMR001) has received CE mark (european conformity in the extended Single Market in the European Economic Area) approval in March 2021. We plan to compare High-Res-OCT as an imaging modality to conventional imaging modalities used in clinical routine, such as the Spectral-Domain-OCT (SD-OCT)

ELIGIBILITY:
Inclusion Criteria:

* Patients from the Department of Ophthalmology, University Hospital Bern requiring conventional imaging for eye disease and willing to sign informed consent Patients of 18 years or older

Exclusion Criteria:

* Patients not willing or able to sign informed consent
* Patients younger than 18 years
* Patients with epilepsy.
* Vulnerable subjects (except the objectives of the investigation concern vulnerable subjects specifically),
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* Enrolment of the PI, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a history of clinically diagnosed ocular disorders, including but not limited to diabetic retinopathy, artery and vein occlusion, glaucoma, optic nerve neuropathy, hereditary retinal diseases/dystrophies, retinal detachment, age related macular degeneration, retinal changes from arterial hypertension, uveitis and healthy individuals undergoing ophthalmic Imaging in Routine clinical practice will be included
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the sensitivity and specificity of High-Res-OCT for retinal fluid | 2 years
  The primary objective of this observational study is to evaluate the sensitivity and specificity to diagnose retinal morphological abnormalities with High-Resolution OCT compared to conventional imaging method (SD-OCT). The main parameter that will be assessed is the presence/absence of retinal fluid. The incidence (binary) of retinal fluid will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT)

SECONDARY OUTCOMES:
Evaluation of the sensitivity and specificity of High-Res-OCT for atrophy area | 2 years
  The incidence (binary) of atrophy area, defined as hypertransmission due to loss of outer retinal layers within the choroidea, will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT)
Evaluation of the sensitivity and specificity of High-Res-OCT for epiretinal membrane | 2 years
  The incidence (binary) of epiretinal membrane (defined as thickening of the retinal nerve fiber layer) will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT)
Evaluation of the sensitivity and specificity of High-Res-OCT for drusen | 2 years
  The incidence (binary) of drusen will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Drusen are defined as hyperfluorescent deposits between the RPE and Bruch's membrane (BM). May be "hard" (small hyperreflective deposits in the retina) and "soft" (larger with indistinct edges).
Evaluation of the sensitivity and specificity of High-Res-OCT for ischemia | 2 years
  The incidence (binary) of ischemia will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Ischemia is defined as hyperreflective band located within/above the outer plexiform layer.
Evaluation of the sensitivity and specificity of High-Res-OCT for neovascularisation | 2 years
  The incidence (binary) of neovascularisation will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Neovascularisation is defined as abnormal growth of vessels from the choroid to the retina through the BM.
Evaluation of the sensitivity and specificity of High-Res-OCT for optic disc swelling | 2 years
  The incidence (binary) of optic disc swelling will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Optic disc swelling is defined as an elevation of the whole nerve head, measured as follows: max. horizontal extent in micrometer of the RNFL (3 mm diameter peripapillary).
Evaluation of the sensitivity and specificity of High-Res-OCT for hyperreflective foci | 2 years
  The incidence (binary) of hyperreflective foci will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Hyperreflective foci are defined as intraretinal hyperreflective dots.
Evaluation of the sensitivity and specificity of High-Res-OCT for scars | 2 years
  The incidence (binary) of scars will be assessed in High-Resolution OCT and compared to conventional imaging method, such as standard-OCT (SD-OCT). Scars are defined as hyperreflective fibrous tissue, which obscures RPE and choroid.
Evaluation of the inter-reader reproducibility | 2 years
  Evaluation of the inter-reader reproducibility of the diagnosis of retinal diseases with High-Res-OCT. Inter-reader reproducibility will be estimated using the Bland-Altman method and the coefficient of repeatability (CoR).
Subgroup analysis | 2 years
  Subgroup analysis will be performed with patients suffering from diabetic retinopathy, artery and vein occlusion, retinal detachment, glaucoma, optic nerve neuropathy, hereditary retinal diseases, age related macular degeneration, retinal changes from arterial hypertension and uveitis. For this purpose, the presence/absence of each above-mentioned morphological abnormality will be assessed/measured in each subgroup and compared with the standard OCT.
Evaluation of the segmentation quality of the retinal layers using High-Res-OCT | 2 years
  For this purpose the discrimination capacity between the different retinal layers will be assessed, i.e. internal limiting membrane, retinal nerve fiber layer, ganglion cell layer, inner plexiform layer, inner nuclear layer, outer plexiform layer, outer nuclear layer, external limiting membrane, photoreceptor layers, retinal pigment epithelium, Bruch's membrane, choriocapillaris, choroidal stroma. For this purpose, a binary outcome will also result, which means that the ability to discriminate between the above-mentioned adjacent layers will be indicated by yes/no.

OTHER OUTCOMES:
Correlation of pathological changes with fundus color photographs | 2 years
  Evaluation whether pathological changes seen in color fundus photography correlate with changes seen in High-Res-OCT. Here, a binary readout, i.e pathology present (yes/no) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Habra, MD, Study Chair — Department of Ophthalmology, University hospital Bern
Locations (1):
- Department of Ophthalmology, Bern University Hospital, Bern, 3010 Bern, Switzerland, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Huang D, Swanson EA, Lin CP, Schuman JS, Stinson WG, Chang W, Hee MR, Flotte T, Gregory K, Puliafito CA, et al. Optical coherence tomography. Science. 1991 Nov 22;254(5035):1178-81. doi: 10.1126/science.1957169.
- [Background] Ly A, Phu J, Katalinic P, Kalloniatis M. An evidence-based approach to the routine use of optical coherence tomography. Clin Exp Optom. 2019 May;102(3):242-259. doi: 10.1111/cxo.12847. Epub 2018 Dec 17. PMID 30560558
- [Background] Guyatt G, Jaeschke R, Heddle N, Cook D, Shannon H, Walter S. Basic statistics for clinicians: 1. Hypothesis testing. CMAJ. 1995 Jan 1;152(1):27-32. PMID 7804919
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Background] de Boer JF, Cense B, Park BH, Pierce MC, Tearney GJ, Bouma BE. Improved signal-to-noise ratio in spectral-domain compared with time-domain optical coherence tomography. Opt Lett. 2003 Nov 1;28(21):2067-9. doi: 10.1364/ol.28.002067. PMID 14587817
- [Background] Bille JF, editor. High Resolution Imaging in Microscopy and Ophthalmology: New Frontiers in Biomedical Optics [Internet]. Cham (CH): Springer; 2019. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK554051/ PMID 32091677
- [Background] Liu YZ, South FA, Xu Y, Carney PS, Boppart SA. Computational optical coherence tomography [Invited]. Biomed Opt Express. 2017 Feb 16;8(3):1549-1574. doi: 10.1364/BOE.8.001549. eCollection 2017 Mar 1. PMID 28663849
- [Background] Wojtkowski M, Srinivasan V, Ko T, Fujimoto J, Kowalczyk A, Duker J. Ultrahigh-resolution, high-speed, Fourier domain optical coherence tomography and methods for dispersion compensation. Opt Express. 2004 May 31;12(11):2404-22. doi: 10.1364/opex.12.002404. PMID 19475077
- [Background] Chen Y, Vuong LN, Liu J, Ho J, Srinivasan VJ, Gorczynska I, Witkin AJ, Duker JS, Schuman J, Fujimoto JG. Three-dimensional ultrahigh resolution optical coherence tomography imaging of age-related macular degeneration. Opt Express. 2009 Mar 2;17(5):4046-60. doi: 10.1364/oe.17.004046. PMID 19259245
- [Background] Ishida S, Nishizawa N. Quantitative comparison of contrast and imaging depth of ultrahigh-resolution optical coherence tomography images in 800-1700 nm wavelength region. Biomed Opt Express. 2012 Feb 1;3(2):282-94. doi: 10.1364/BOE.3.000282. Epub 2012 Jan 11. PMID 22312581
- [Background] An L, Li P, Shen TT, Wang R. High speed spectral domain optical coherence tomography for retinal imaging at 500,000 A-lines per second. Biomed Opt Express. 2011 Oct 1;2(10):2770-83. doi: 10.1364/BOE.2.002770. Epub 2011 Sep 12. PMID 22025983
- [Background] Tsang SH, Sharma T. Fluorescein Angiography. Adv Exp Med Biol. 2018;1085:7-10. doi: 10.1007/978-3-319-95046-4_2. PMID 30578475
- [Background] Mitchell P, Liew G, Gopinath B, Wong TY. Age-related macular degeneration. Lancet. 2018 Sep 29;392(10153):1147-1159. doi: 10.1016/S0140-6736(18)31550-2. PMID 30303083
- [Background] Ferris FL, Davis MD, Clemons TE, Lee LY, Chew EY, Lindblad AS, Milton RC, Bressler SB, Klein R; Age-Related Eye Disease Study (AREDS) Research Group. A simplified severity scale for age-related macular degeneration: AREDS Report No. 18. Arch Ophthalmol. 2005 Nov;123(11):1570-4. doi: 10.1001/archopht.123.11.1570. PMID 16286620
- [Background] Wolf S, Wolf-Schnurrbusch U. Spectral-domain optical coherence tomography use in macular diseases: a review. Ophthalmologica. 2010;224(6):333-40. doi: 10.1159/000313814. Epub 2010 May 4. PMID 20453539
- [Background] Saito T, Rehmsmeier M. The precision-recall plot is more informative than the ROC plot when evaluating binary classifiers on imbalanced datasets. PLoS One. 2015 Mar 4;10(3):e0118432. doi: 10.1371/journal.pone.0118432. eCollection 2015. PMID 25738806

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT05130385/Prot_SAP_000.pdf